CLINICAL TRIAL: NCT04379479
Title: Assessment of the Clinical Effect of Dialyzable Leukocyte Extracts in Individuals With Acute Respiratory Infection (Suspected or Confirmed Cases of COVID-19) (FUTURE-T)
Brief Title: Clinical Effect of Dialyzable Leukocyte Extract in Suspected or Confirmed Cases of COVID-19 (FUTURE-T)
Acronym: FUTURE-T
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Polytechnic Institute, Mexico (Other)
Responsible Party: Principal Investigator, Toni Homberg von Thaden, Principal Investigator, National Polytechnic Institute, Mexico
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IC-20-001; SH-001-2020 (Other: Instituto Politécnico Nacional)
Record Dates: First submitted 2020-05-01; First posted 2020-05-07 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: COVID-19; SARS-CoV-2 Infection
Keywords: Dialyzable leukocyte extract; Treatment COVID-19; Treatment SARS-CoV-2 infection
MeSH Terms: conditions — COVID-19 | interventions — Transfer Factor

STUDY DESIGN:
Intervention Model Description: Exploratory clinical trial, prospective, longitudinal, placebo-controlled, double-blinded, in patients with symptoms of non-severe acute respiratory infection (suspected/confirmed cases of COVID-19).
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dialyzable Leukocyte Extract (Experimental): Oral administration 2 mg/5 mL every 24 hours for 14 days, following by 2 mg/5 mL twice a week for 3 weeks.
  All patients will receive paracetamol as symptomatic treatment, 500 mg oral administration 3 times per day.
  Interventions: Drug: Dialyzable Leukocyte Extract
- Placebo (Placebo Comparator): Oral administration 5 mL every 24 hours for 14 days, following by 5 mL twice a week for 3 weeks.
  All patients will receive paracetamol as symptomatic treatment, 500 mg oral administration 3 times per day.
  Interventions: Drug: Placebo oral

INTERVENTIONS:
Drug: Dialyzable Leukocyte Extract — Experimental Intervention. Dialyzable Leukocyte Extract
  Other Names: Transferon oral
  Arms: Dialyzable Leukocyte Extract
Drug: Placebo oral — Placebo
  Other Names: Placebo comparator
  Arms: Placebo

SUMMARY:
Main goal: To generate information on the efficacy and safety of Dialyzable Leukocyte Extract (DLE) as an aid in the treatment of patients with acute respiratory infection (suspected or confirmed cases of COVID-19).

Primary goal: To generate information on the efficacy of DLE as an aid in symptomatic treatment, by reducing the signs and symptoms of acute respiratory infection (suspected/confirmed cases of COVID-19).

Secondary goals:

1. To evaluate clinical deterioration and respiratory alarm data.
2. To evaluate the duration of the clinical picture.
3. To explore cytokine changes associated with the therapeutic effect induced by DLE.
4. To obtain data on the safety of DLE as an aid in the symptomatic treatment of acute respiratory infection (suspected/confirmed cases of COVID-19).
5. To generate information to validate the contingency scale to assess the severity of acute respiratory disease (suspected/confirmed cases of COVID-19).

Justification The systemic inflammatory response has been recognized as being responsible for COVID-19 complications. Immunomodulation strategies to control it are currently being considered, including the use of systemic steroids to down-regulate the systemic inflammatory response, the use of human immunoglobulin and even chloroquine given its anti-inflammatory and antiviral qualities; however, none of these treatments has been sufficiently studied or has shown any significant change in the clinical course of infected patients.

Due to the importance of the COVID-19 pandemic and in the absence of specific treatment, it is important to implement new treatments that allow modulating the immune response, and one strategy may be the addition of DLE to symptomatic and supportive treatment.

Hypotheses by goals.

1. The addition of DLE to the symptomatic treatment could decrease the severity of the clinical outcome (signs and symptoms) in individuals with an acute respiratory infection (cases suspected/confirmed by COVID-19).
2. The addition of DLE to the symptomatic treatment could decrease the clinical deterioration due to the acute respiratory infectious process (suspected/confirmed cases of COVID-19).
3. The addition of DLE to the symptomatic treatment could decrease the duration of the clinical outcome (suspected/confirmed cases of COVID-19).

DETAILED DESCRIPTION:
Dialyzable Leukocyte Extract (DLE) (Transferon oral®) is a dialyzed extract obtained from human leukocytes. Its active ingredient is a complex mixture of low molecular weight peptides obtained from dialysis (12 kDa), and subsequent ultrafiltration (10 kDa) of lysed leukocyte and platelet concentrates. This product is manufactured by Laboratory of Scientific Research (Pharma-FT) at the Nacional School of Biological Sciences (ENCB), National Polytechnic Institute (IPN) using a patented method in Mexico (MX/a/2011/013852), USA (US9328152B2), EU (EPA-126128), Canada (2860260), Peru (000969-2014/DIN) and Colombia (14138326).

DLE is a complex drug, the active principle is multiple peptide units. Thus, DLE cannot be fully characterized, requiring the application of analytical techniques that can describe the overall behavior of all of its components (peptide polydispersity).

Two orthogonal techniques have been used to determine the molecular weight of the peptide components of DLE based on their migration through a polymer matrix. The molecular weight of 10 kDa was determined by polyacrylamide gels electrophoresis under denaturing conditions (SDS-PAGE), while a molecular weight lower than 15 kDa was determined by molecular exclusion chromatography.

The peptide nature of DLE has been demonstrated using an aminogram method. This method includes the acidic hydrolysis of the peptide components until free amino acids are obtained, which are derivatized and identified based on the retention time of an amino acid standard using reverse phase chromatography (RP-UPLC). Additionally, the peptides of this drug were determined to be highly soluble by RP-UPLC coupled to UV, while mass spectometry, coupled to RP-UPLC, exhibited consistent ionization patterns.

Non-clinical and clinical studies relevant to this research. Experimentally, in a murine model of virus infection, administration of DLE showed a decrease in serum concentrations for TNF and IL-6, accompanied by an increase of IFN. In humans, viral etiology is responsible for 90-95% of cases of respiratory tract infections. The common viruses involved in respiratory diseases are rhinoviruses (∼50%), coronaviruses (∼10%), adenoviruses, respiratory syncytial virus, influenza, and parainfluenza viruses (which generally add up between 10% to 15%), human metapneumovirus (<5 %). The first evidence that DLE might have a therapeutic effect in respiratory infections arose from the analysis of a series of cases (36 adults and 63 children) with allergic rhinitis who received DLE in addition to the standard treatment. 11% of adults and 25.4% of children reported a decrease in the frequency of respiratory infections. Similarly, in a series of 70 adults and 54 children with persistent moderate asthma who received treatment with DLE as adjuvant therapy, 44% of adults and 31% of children reported a decrease in the frequency of respiratory infections, in addition to the improvement of allergic symptoms. In a study of 52 individuals, the effectiveness of DLE was evaluated by reducing the severity and frequency of infectious symptoms. That study showed a decrease in the frequency and in the severity of the infectious respiratory symptoms (77.1%) in pediatric patients. In comparison, 82.4% of adults decrease the frequency and/or diminish the severity of infectious respiratory symptoms. In a clinical follow-up of pediatric patients with sepsis to whom DLE was added to the standard treatment decrease in C-reactive protein levels, reduction in the neutrophil count at 72 hours after hospitalization, and an increase in the survival rate of 30% was reported.

SARS-CoV-2 induces significant lung damage due to uncontrolled and dysregulated inflammatory activity, then immunomodulatory drugs have been suggested as treatment. The findings related to DLE, support their immunomodulatory capacity as a potential therapeutic tool in infectious respiratory diseases with a prominent inflammatory component.

Primary goal. To generate information on the efficacy of DLE as an aid in symptomatic treatment, by reducing the signs and symptoms of acute respiratory infection (suspected/confirmed cases of COVID-19).

Secondary goals.

1. To evaluate clinical deterioration and respiratory alarm data.
2. To assess the duration of the clinical manifestations.
3. To explore cytokine changes
4. To obtain data on the safety of DLE as an aid in the symptomatic treatment of acute respiratory infection (suspected/confirmed cases of COVID-19).
5. To generate information to validate the contingency scale (CS) to assess the severity of acute respiratory disease (suspected/confirmed cases of COVID-19).

Hypothesis. The addition of DLE to the symptomatic treatment will reduce the signs and symptoms of acute respiratory infection.

The recruitment method will be achieved electronically.

The acute respiratory infection will be classified according to its clinical symptoms, following the Mexican Clinical Guideline in which COVID-19 disease is divided into non-serious and severe cases. The clinical evaluation of the patient will be assessed by a CS designed for this study, and includes three major items subdivided into minor items (range 0 to 4 in each one):

General symptoms: Fever, Headache Superior airway respiratory symptoms: Sneezing, nasal congestion, runny nose Lower airway respiratory symptoms: Cough, Dyspnea, and Pain or Sense of constriction or oppression in the chest.

Statistics. Four populations will be considered for the analysis: randomized individuals in the study or full analysis set (FAS), safety population (SP), the population of the intention-to-treat (ITT), and population per-protocol (PP).

The FAS population will consist of all individuals who were randomized into the study (they are assigned a random number). The ITT population will consist of all patients who were randomized, who received at least one dose of the study drug, and who had at least one assessment of the primary or secondary endpoints after the baseline assessment. Following the principle of the intention of treatment, patients will be analyzed according to the treatment assigned during randomization. The SP will consist of all patients who received at least one dose of the study drug and who have at least one safety assessment after the baseline assessment. The patients will be analyzed according to the treatment they received. As a clarifying note, the statement that the patient has no adverse events constitutes a safety assessment. The PP will consist of all patients in the ITT population who complete all visits, who have an accurate evaluation of the primary efficacy variable, and who do not contain significant protocol violations.

Statistical methods. Demographic data, clinical history, and key baseline efficacy variables for all randomized patients will be summarized by treatment group in tables (number and percentage) for qualitative variables; and in tables containing the average, standard deviation, median, minimum and maximum, by treatment group, for the quantitative variables. A comparison of groups at the baseline visit will be analyzed using Chi-square tests for qualitative variables and two-sample student t-tests for quantitative variables (p-values will be provided for descriptive purposes only). Additionally, the medical history, concomitant medications, comorbidities will be summarized using frequency tables.

Primary outcome. The primary result of efficacy will be the measurement of the score of the CS at the end of treatment or early termination, in the ITT population. The algorithm of the imputation of the last observation carried forward (LOCF) will be applied in the case of patients who withdraw, discontinue therapy, or withdraw from the study. The primary analysis will be performed using the ITT population. This analysis will also be performed in the PP population to assess the robustness of the results. The primary outcome will be analyzed with a covariance model that includes the treatment group, baseline value, and center.

The exploratory hypothesis of the primary objective is to establish whether there could be a difference in the decrease in the score of the CS at the end of treatment, under a superiority hypothesis approach described below:

Ho: µPlacebo - µDLE>0 Ha: µPlacebo - µDLE<0

Possible superiority of the DLE addition as an aid to symptomatic treatment relative to symptomatic/placebo treatment will be established if the upper limit of the 2-sided 95% confidence interval for the difference µPlacebo-µDLE is less than 0.

Secondary outcomes. The appearance of respiratory alarm data will be identified in the study groups, presenting the results in a frequency chart with the proportion of patients who presented alarm data by group. It will be analyzed using the Chi-Square test. The duration of clinical manifestations corresponds to the number of days with any of the signs and symptoms described in the CS. Descriptive statistics will be performed in each treatment group; the comparison will be made using the student's t-test. Immunological changes are defined as changes in the total leukocyte count, total lymphocytes, ESR, and serum concentration of CRP, procalcitonin, D-dimer, ferritin, CK, myoglobin, IL-6, TNF, interferons, and specific antibodies for the virus. Descriptive statistics will be presented by treatment group vs. visit, as well as the proportion of patients who show normalization of values during treatment.

Sample size. Due to the lack of information on the efficacy of the study drug in cases of acute respiratory infection with COVID-19, the statistical calculation of the sample size does not apply. However, as a descriptive exercise, given the current contingency by COVID-19 pandemic, an estimation of the sample size is proposed in this study based on the CS that has been specifically designed for this study. Contingency score ranges from 0 to 32, considering that the study population is non-severe patients, the scoring average will correspond to the order of 16 points with a standard deviation of 4. It has also been assumed that the scoring behavior is that of a continuous variable with a normal distribution.

The sample size calculation procedure is by means of the Julious 2004/FARTSSIE22 equation for superiority designs in parallel with two groups (DLE vs. Placebo). According to the following values:

a. Type I error: 0.05 (5%); b. Type II error: 0.2 (20%). Power: 1-b: 0.8 (80%) Proposed standard deviation: 4 Difference to detect between groups: 1 The sample size relationship between groups: 1:1 (balanced) The sample size calculated is 253 per group. An additional 10% (q) will be included to offset withdrawals from the study or treatment; therefore, 562 patients (nt) 281 will be randomized by treatment in order to have the estimated number of patients for the hypothesis test. nt=n/1-q =506/0.9=562

Procedures to explain missing data. Missing data for the variables that are measured on a single occasion cannot be substituted, and that individual cannot be included in the analysis. For data that is measured on more than one time, in case of missing data, the last value measured after the baseline will be taken into account. (LOCF)

Procedures for reporting any deviation from the statistical plan. If there are deviations from the original statistical plan, these will be described and justified in the final report.

Selection of individuals to be included in the analysis. All randomized individuals who have received at least one dose of the investigational product under the maxim of ITT will be included in the analysis.

Access to information. The study will be monitored by specific personnel; internal and external inspections and audits will be allowed and facilitated, allowing access to information while maintaining the confidentiality of the study individuals.

ELIGIBILITY:
Inclusion Criteria:

1. Adults who agree to participate and sign informed consent.
2. Suspected case, according to the operational definition (CONAVE).*
3. In the case of confirmed cases, will be those individuals who meet the operational definition of a suspected case and have a confirmed diagnosis by molecular biology, according to the operational definition (CONAVE).**
4. The time of acute respiratory symptoms should be no longer than 72h.
5. Negative to the rapid test for influenza A/B.
6. Live in an urban area with easy access for visits.

   * Person of any age that has presented at least two of the following signs and symptoms: cough, fever or headache

Accompanied by at least one of the following signs or symptoms:

Dyspnea (signal of severity) Arthralgia Myalgia Odynophagia / pharyngeal burning Rhinorrhea Conjunctivitis Chest pain

**SARS-CoV2 infection confirmed by molecular diagnostic by one laboratory from the National Network of Public Health Laboratories recognized by InDRE.

Exclusion Criteria:

1. Pregnancy.
2. Evidence of severe acute respiratory infection, even if it meets the criteria for a suspected or confirmed case.
3. Hepatic insufficiency
4. Diseases that occur with immunosuppression or therapeutic immunosuppression.
5. Heart diseases; controlled hypertension is allowed.
6. Metabolic diseases; controlled diabetes mellitus is allowed.
7. Individuals who have been treated with DLE in the last 6 months.

CONAVE: National Committee for Epidemiological Surveillance. InDRE: Institute of Epidemiological Diagnosis and Reference.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 562 (Estimated)
Dates: Start 2020-05 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Change in the score of the "Contingency scale to assess the severity of acute respiratory disease in cases suspected/confirmed by COVID-19" | 35 days
  Change in the score of the "Contingency scale to assess the severity of acute respiratory disease in cases suspected/confirmed by COVID-19" at the end of treatment concerning the baseline value. The clinical effect will be daily evaluated with the patient's diary in the cell app. Minimum value 0, Maximum value 32 points. Higher scores mean worse outcome.

SECONDARY OUTCOMES:
Clinical deterioration | 35 days
  Defined as the presence of signs and symptoms related with respiratory alarm symptoms. The respiratory alarm data will be daily evaluated with the patient's diary in the cell app.
Duration of the clinical status | 35 days
  Defined as the number of days with any of the symptoms mentioned in contingency table during the visits and follow-up through the patient's diary in the cell app.

OTHER OUTCOMES:
Cytokine concentration | 35 days
  Defined as the changes in the total concentration of the serum cytokines IL-6, TNF-α and type I and II Interferons due to DLE treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Mayra Pérez-Tapia, PhD, Study Director — Instituto Politecnico Nacional; Maria C Jimenez-Martínez, MD PhD, Study Director — Universidad Nacional Autonoma de Mexico; Toni A Homberg von Thaden, MD, Principal Investigator — National Polytechnic Institute, Mexico
Locations (1):
- Escuela Nacional de Ciencias Biológicas, Instituto Politécnico Nacional, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
All data will be shared that underlies results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will become available immediately at the end of study.
Access Criteria: All data will be published in a scientific journal.

REFERENCES:
- [Background] Carballo-Uicab G, Linares-Trejo JE, Mellado-Sanchez G, Lopez-Morales CA, Velasco-Velazquez M, Pavon L, Estrada-Parra S, Perez-Tapia SM, Medina-Rivero E. Validation of a Cell Proliferation Assay to Assess the Potency of a Dialyzable Leukocyte Extract Intended for Batch Release. Molecules. 2019 Sep 20;24(19):3426. doi: 10.3390/molecules24193426. PMID 31547184
- [Background] Avila S, Munoz-Garcia L, Vazquez-Leyva S, Salinas-Jazmin N, Medina-Rivero E, Pavon L, Mellado-Sanchez G, Chacon-Salinas R, Estrada-Parra S, Vallejo-Castillo L, Perez-Tapia SM. Transferon, a peptide mixture with immunomodulatory properties is not immunogenic when administered with various adjuvants. J Immunotoxicol. 2017 Dec;14(1):169-177. doi: 10.1080/1547691X.2017.1346009. PMID 28707490
- [Background] Ramirez-Ramirez D, Vadillo E, Arriaga-Pizano LA, Mayani H, Estrada-Parra S, Velasco-Velazquez MA, Perez-Tapia SM, Pelayo R. Early Differentiation of Human CD11c+NK Cells with gammadelta T Cell Activation Properties Is Promoted by Dialyzable Leukocyte Extracts. J Immunol Res. 2016;2016:4097642. doi: 10.1155/2016/4097642. Epub 2016 Oct 25. PMID 27847830
- [Background] Medina-Rivero E, Vallejo-Castillo L, Vazquez-Leyva S, Perez-Sanchez G, Favari L, Velasco-Velazquez M, Estrada-Parra S, Pavon L, Perez-Tapia SM. Physicochemical Characteristics of Transferon Batches. Biomed Res Int. 2016;2016:7935181. doi: 10.1155/2016/7935181. Epub 2016 Jul 20. PMID 27525277
- [Background] Salinas-Jazmin N, Estrada-Parra S, Becerril-Garcia MA, Limon-Flores AY, Vazquez-Leyva S, Medina-Rivero E, Pavon L, Velasco-Velazquez MA, Perez-Tapia SM. Herpes murine model as a biological assay to test dialyzable leukocyte extracts activity. J Immunol Res. 2015;2015:146305. doi: 10.1155/2015/146305. Epub 2015 Apr 23. PMID 25984538
- [Background] Medina-Rivero E, Merchand-Reyes G, Pavon L, Vazquez-Leyva S, Perez-Sanchez G, Salinas-Jazmin N, Estrada-Parra S, Velasco-Velazquez M, Perez-Tapia SM. Batch-to-batch reproducibility of Transferon. J Pharm Biomed Anal. 2014 Jan;88:289-94. doi: 10.1016/j.jpba.2013.09.004. Epub 2013 Sep 17. PMID 24099727
- [Background] Homberg T, Sáenz V, Galicia-Carreón J, Lara I, Cervantes-Trujano E, Andaluz MC, Vera E, Pineda O, Ayala-Balboa J, Estrada-García A, Estrada-Parra S, Pérez-Tapia M, Jiménez-Martínez MC.The adverse event profile in patients treated with Transferon TM (Dialyzable leukocyte extracts): A preliminary report. Pharmacology & Pharmacy. 2015; 6(02): 65.
- See also: Official site — https://www.encb.ipn.mx